CLINICAL TRIAL: NCT07363577
Title: A Randomized, Double-blinded, Placebo-controlled, Multicenter Study to Evaluate the Antipsychotic Efficacy and Safety of LB 102 in the Treatment of Adult Patients With Acute Schizophrenia
Brief Title: Study to Evaluate LB-102 for the Treatment of Adult Patients With Acute Schizophrenia
Acronym: NOVA2
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: LB Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LB-102-008
Record Dates: First submitted 2025-12-26; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia
Keywords: acute schizophrenia,; exacerbated acute schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Tablets

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1:1 to one of three treatments
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LB-102 (50 mg tablet) (Experimental): • LB-102 50 mg given orally for 6 weeks
  Interventions: Drug: LB-102 (50 mg tablet)
- LB-102 (100 mg tablet) (Experimental): LB-102 100 mg given orally for 6 weeks
  Interventions: Drug: LB-102 (100 mg tablet)
- Placebo (Placebo Comparator): Placebo given orally for 6 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: LB-102 (50 mg tablet) — LB-102 oral tablet given for six weeks
  Other Names: LB-102
  Arms: LB-102 (50 mg tablet)
Drug: LB-102 (100 mg tablet) — LB-102 oral tablet given for six weeks
  Other Names: LB-102
  Arms: LB-102 (100 mg tablet)
Other: Placebo — Placebo tablet given orally for six weeks
  Arms: Placebo

SUMMARY:
This is a Phase 3, randomized, double blind, placebo controlled, fixed dose, study designed to evaluate the efficacy, safety, tolerability, and of LB-102 versus placebo for the treatment of adult patients with an acute exacerbation of schizophrenia.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double blind, placebo controlled, fixed dose, multicenter study designed to assess the efficacy, safety, tolerability, and pharmacokinetics (PK) of LB-102 100 mg once daily (QD) and LB-102 50 mg QD versus placebo QD for the treatment of adult patients with an acute exacerbation of schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* Able to provide ICF
* Willing to be hospitalized for duration of the study
* Diagnosis of schizophrenia as defined by DSM-5
* BMI - 18-40
* PANSS 80-120

Exclusion Criteria:

* Sexually active m/f not willing to adhere to highly effect birth control
* Breast feeding
* Increase in PANSS of > 20% between screening and baseline
* History of resistant treatment to schizophrenia medications
* DSM-5 diagnosis other than schizophrenia
* Risk of suicidal behavior
* Risk of violent or destructive behavior
* Clinically significant tardive dyskinesia determined by a score of ≥3 on Item 8 of the AIMS at Screening
* Score of ≥3 on the BARS global clinical assessment of akathisia at Screening
* Insulin dependent diabetes
* Known ischemic heart disease or any history of myocardial infarction, congestive heart failure (whether controlled or uncontrolled), angioplasty, stenting, or coronary artery bypass surgery
* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or oncologic disease or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the patient

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to Week 6 on the Positive and Negative Syndrome Scale | 6 weeks
  Determine whether LB-102, demonstrates antipsychotic efficacy, as determined by a change from Baseline on the Positive and Negative Syndrome Scale (PANSS) total score, compared to placebo: increase in scale indicates worsening while a decrease in the scale likely indicates a response to treatment

SECONDARY OUTCOMES:
Evaluate the Safety and Tolerability of LB-102 | 10 weeks
  Evaluate the safety and tolerability of LB-102 in patients by evaluating adverse events
Change in Clinical Global Impressions-Severity of Illness scale (CGI-S) | 6 weeks
  Assess the effect of LB-102 on the treatment for schizophrenia, as determined by a change from Baseline in the Clinical Global Impressions Severity of Illness scale: whereas increase demonstrates worsening of illness and decrease in score likely indicates response to treatment

CONTACTS AND LOCATIONS:
Overall Officials: John Kane, MD, Principal Investigator — Northwell Health

IPD SHARING:
Plan to Share IPD: No